CLINICAL TRIAL: NCT03856281
Title: Intermittent Pneumatic Compression for Treating Lower Limb Lymphoedema (IMPRESS II)
Brief Title: Intermittent Pneumatic Compression for Treating Lower Limb Lymphoedema
Acronym: IMPRESS II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cwm Taf University Health Board (NHS) (Other Government)
Collaborators: University of South Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPRESS II
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-02

CONDITIONS: Lymphoedema of Leg
MeSH Terms: interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group A (Experimental): LymphAssist IPC device - participants act as their own control for 5 weeks, receiving standard care only. After 5 weeks the group use the device twice a day, every day for a 5 week period.
  Interventions: Device: Intermittent Pneumatic Compression
- Intervention Group B (Experimental): Sequential IPC device - participants act as their own control for 5 weeks, receiving standard care only. After 5 weeks the group use the device twice a day, every day for a 5 week period.
  Interventions: Device: Intermittent Pneumatic Compression

INTERVENTIONS:
Device: Intermittent Pneumatic Compression — Participants administer an intermittent pneumatic compression device in addition to their standard lymphoedema care for a 5 week treatment period
  Other Names: LymphAssist

SUMMARY:
The treatment of lymphoedema and its associated complications represent a considerable drain on increasingly limited NHS resources. Intermittent pneumatic compression (IPC) represents an innovative treatment for this condition, however the efficacy of IPC as a treatment for lower limb lymphoedema needs to be investigated via robust clinical research.

DETAILED DESCRIPTION:
The primary aim of this research is to evaluate the effectiveness of intermittent pneumatic compression (IPC) as a treatment for lower limb lymphoedema as a whole, and to compare the effectiveness of a new generation device, in this case the LymphAssist (Huntleigh Healthcare), against older sequential models. The study methodology consists of a pilot randomised control trial of two groups - Intervention group A will continue to receive their standard lymphoedema care but will also be provided with a LymphAssist IPC device to use, mimicking manual lymph drainage therapy. Participants in intervention group B will receive their standard care plus an IPC device that uses sequential therapy. Each participant will act as a control for a 5 week period continuing with their standard treatment only. Outcome measures include impact on limb volume, skin stiffness and elasticity score and impact on quality of life scores.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over,
* Able to provide written consent,
* Confirmed diagnosis of lower limb ISL stage II or III.

Exclusion Criteria:

* • Unable to provide written consent

  * Severe congestive heart failure
  * Severe skin problems, lower limb ulcers or wounds.
  * Presence of cognitive impairment (permanent or intermittent) which would prevent patients from using the IPC device safely or adhering to instructions/study protocol.
  * Non-pitting chronic lymphoedema.
  * Known or suspected deep vein thrombosis.
  * Pulmonary embolism.
  * Thrombophlebitis.
  * Acute inflammation of the skin (erysipelas, cellulitis).
  * Uncontrolled/severe cardiac failure.
  * Pulmonary oedema.
  * Ischaemic vascular disease.
  * Active cancer diagnosis.
  * Active metastatic diseases affecting the oedematous region.
  * Oedema at the root of the extremity or truncal oedema.
  * Severe peripheral neuropathy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Leg Volume | 5 weeks
  Circumferential measurements at every 4cm from the top of the ankle to the thigh will be used to calculate limb volume in mls

SECONDARY OUTCOMES:
Myoton Scores | 5 weeks
  The effect IPC has on skin stiffness (N/m), tone (Hz) and elasticity (D)
Quality of Life Scores | 5 weeks
  The effect IPC has on quality of life scores - raw score created from a series of Likert Scales

CONTACTS AND LOCATIONS:
Overall Officials: Mark Williams, PhD, Principal Investigator — University of South Wales
Locations (1):
- Dewi Sant Hospital, Pontypridd, United Kingdom

IPD SHARING:
Plan to Share IPD: No